CLINICAL TRIAL: NCT03876093
Title: Epilepsy-related Brain Tumors Register
Status: Withdrawn | Type: Observational
Why Stopped: The PI decided.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Epilepsy-related brain tumors
Record Dates: First submitted 2019-03-07; First posted 2019-03-15 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epilepsy is defined by a cerebral disorder characterized by a lasting predisposition to generate epileptic seizures and by the neurobiological, cognitive, psychological and social consequences of this affection. The definition of epilepsy requires the occurrence of at least one epileptic seizure. 1% of the population suffers from epilepsy. The most common causes are genetic and vascular, 10% of epileptic syndromes are caused by a tumor.

The incidence of brain tumors in people with epilepsy is approximately 4%. Among patients with brain tumor (s), the frequency of epilepsy is 30% or more depending on type of tumeur. 30-50% of brain tumors are revealed by an epileptic seizure and 10 to 30% of patients with brain tumor (s) will develop seizures during their evolution.

The main objective is to evaluate the frequency of epileptic seizures according to the type of brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* patient whose age ≥ 18 years
* Patient hospitalized or seen in consultation in the Department of Neurology within the Hospital Group Paris Saint-Joseph
* Diagnosis of primary or secondary brain tumor, radiologically and / or histologically
* Epilepsy revealing or occurring in a patient developing a brain tumor
* Francophone patient

Exclusion Criteria:

* Pre-existing and known epilepsy before the diagnosis of brain tumors
* Epilepsy occurring within 2 weeks postoperatively
* Anteriority of taking antiepileptic treatment
* Patient under tutorship or curatorship
* Patient deprived of liberty
* Patient with comprehension disorders making it impossible to understand the protocol
* Patient or relative opposing the use of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized following an epileptic seizure or seen in consultation in the neurology department of the GHPSJ, diagnosed with primary or secondary brain tumor from January 2013 to December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
number of epileptic seizures | Day 1
  number of epileptic seizures at the time of neurology consultation or hospitalization

SECONDARY OUTCOMES:
number of epileptic seizures | until 10 years
  number of epileptic seizures at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Roubeau Vincent, MD, Principal Investigator — Fondation Hôpital Saint-Joseph